CLINICAL TRIAL: NCT07209020
Title: Safety Observation of HealiAid Collagen Wound Dressing in Patients Undergoing Breast Tumor Surgery: A Post-Market Clinical Trial
Brief Title: HealiAid Collagen Wound Dressing in Patients Undergoing Breast Tumor Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBI-HAS-202403
Record Dates: First submitted 2025-09-22; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Tumors; Wound Healing; Collagen Wound Dressing
Keywords: breast tumors; wound healing; collagen wound dressing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAS (Experimental)
  Interventions: Device: HealiAid Collagen Wound Dressing

INTERVENTIONS:
Device: HealiAid Collagen Wound Dressing — Within the surgery procedure, the tumor is completely removed and the wounds are cleaned properly before applying the HealiAid Collagen Wound Dressing. HealiAid is soft and pliable. It can be adjusted to the size of the wound, and it is recommended to apply one to four pieces per wound. HealiAid Collagen Wound Dressing will be kept in place until absorbed completely.

SUMMARY:
The goal of this clinical trial is to evaluate the safety of the collagen wound dressing (HealiAid) in breast tumor patients with surgical treatment. The main questions it aims to answer are:

1. To record the incidence of the postoperative complications and adverse events (AEs) after applying the HealiAid wound dressing in patients undergoing surgery for breast tumor.
2. To evaluate the patients' satisfaction and quality of life using the Breast Q questionnaire before surgery and at weeks 2, 12, 26, and 52 after the surgery.
3. To evaluate the patients' results of vital signs, hematology tests, tumor marker tests, breast ultrasonography, and mammography after the surgery.

Participants will undergo a breast surgery. Within the surgery procedure, the tumor will be completely removed with a margin of 1-2 cm surrounding healthy tissue and the wounds will be cleaned properly before the patients receive the HealiAid Collagen Wound Dressing at treatment visit, and six follow up visits at week 1, 2, 4, 12, 26 and 52.

DETAILED DESCRIPTION:
This study is an open label, multicenter post-market clinical follow-up study with a single arm group design. Included patients with confirmed diagnosis of breast tumor who are candidates for surgical treatment, including breast partial mastectomy (BPM), breast conserving surgery (BCS), sentinel lymph node dissection (SLND) and/or axillary lymph node dissection (ALND).

Within the surgery procedure, the tumor is completely removed with a margin of 1-2 cm around healthy tissue. Wounds are then cleaned properly before applying the HealiAid Collagen Wound Dressing. HealiAid is soft and pliable. It can be adjusted to the size of the wound, and it is recommended to apply one to four pieces per wound. HealiAid Collagen Wound Dressing will be kept in place until absorbed completely.

The rehabilitation and the related introduction postoperative will follow the hospital protocols, patients will be advised to mobilize the ipsilateral arm within a few hours after surgery.

Patients will be visited at weeks 1, 2, 4, 12, 26, and 52 after surgery and assessed for surgical site wound and AE assessment. Additionally, photographs of the breast appearance are taken post-surgery before discharge and at weeks 12, and 52 after the surgery. Patient's quality of life (QoL) and satisfaction are evaluated using the Breast-Q questionnaire on screening day, before surgery on day 1, and at weeks 2, 12, 26, and 52 after the surgery.

Vital signs including respiratory rate, pulse, blood pressure and temperature will be continuously measured during the patients' hospitalization period following the surgery, which is estimated to last up to 3 days.

For the follow up examination, the breast ultrasonography will be performed at week 2 and 26 and week 52, and mammography will be performed at week 52. The hematology test and Tumor marker test will be performed at week 26.

All hypothesis tests are two-sided, use α=0.05, if P<0.05, it is considered statistically significant. For inferential statistics, comparison of quantitative data, use the t-test or Wilcoxon rank sum test. For count data comparison, use Chi-square test or Fisher's exact test. For continuous data comparison, use repeated measured ANOVA test. For main/significant safety indicators, consider the influence of center or other stratification factors and perform Pearson correlation test (with baseline data as covariates).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old.
* Patients are diagnosed with a benign or malignant breast tumor, that tumor size of ≦ 5 cm and no distant metastasis assessed by the imaging (breast ultrasonography, mammography, or MRI) and pathologic examination within 12 weeks before screening. If a benign breast tumor is identified through imaging and subsequently removed via surgery performed after the subject's enrollment in the study, the pathology report from that surgery should be used instead of any previous report.
* Patients diagnosed with a breast tumor, or those with a history of radiation and chemotherapy, who are scheduled to undergo surgery such as partial mastectomy, breast-conserving surgery, sentinel lymph node dissection, and/or axillary lymph node dissection .
* Patients who understand and are able to comply with follow-up visits and treatment during the trial period.
* Patients who are willing and capable of providing written informed consent. Not a person subject to a sentence of guardianship or subject to judicial guardians.

Exclusion Criteria:

* Patients with breast cancer stage III or IV.
* Patients with inflammatory breast cancer.
* Patients with multicentric lesions or lesions with diffuse microcalcification.
* Patients with retro areolar breast carcinoma.
* Have a history of severe allergies or are allergic to collagen.
* Collagen vascular disease.
* History of serious postoperative complications.
* Infected wound.
* Patients who require emergency surgery.
* Patients with coagulation dysfunction, such as abnormal preoperative coagulation time (prothrombin time (PT)>18 seconds or partial thromboplastin time (PTT) >50 seconds)
* Patients with untreated or unstable diabetes, that the fasting blood sugar >180 mg/dL or postprandial blood sugar >200 mg/dL.
* Patients with untreated or unstable chronic diseases, such as hypertension, hyperlipidemia, cardiovascular disease, stroke.
* Patients with Body mass index (BMI) > 30.
* Patients who are pregnant or breastfeeding women.
* Patients with drug abuse or addiction.
* Others who have been judged by the principal investigator as participating in this trial will endanger their physical and mental health.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the postoperative complications and adverse events | Day0 through out 52 weeks
  The incidence of the postoperative complications and adverse events (AEs) using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and to assess surgical site wounds after applying the HealiAid wound dressing in patients undergoing surgery for breast tumor.

SECONDARY OUTCOMES:
Satisfaction and quality of life | before surgery and at weeks 2, 12, 26, and 52 after the surgery.
  To evaluate the patients' satisfaction and quality of life using the questionnaire: Breast Q Breast Conserving Therapy Module. Scores range from 0 to 100, with higher scores indicating better satisfaction and quality of life.
Number of participants with abnormal vital sign results | From post-surgery until discharge, assessed up to 3 days.
  Number of participants who present with abnormal vital sign results. Vital signs include respiratory rate, pulse, blood pressure and temperature. The vital sign will be continuously measured post-surgery to discharge, which is estimated to last up to 3 days.
Number of participants with abnormal laboratory tests results | Week 26 after the surgery.
  Number of participants who present with abnormal hematology test result at Week 26. Hematology test including the data of white blood cell (WBC) count, red blood cell (RBC) count, hemoglobin (Hgb), hematocrit (Hct), platelet (PLT) count.
Number of participants with abnormal tumor marker test results | Week 26 after the surgery.
  Number of participants with abnormal tumor marker results for breast cancer including CA-153 and CEA.
Breast ultrasonography | Weeks 2, 26, and 52 after the surgery
  Breast ultrasonography may be postponed to Visit 4 (Week 4 ±7 days) if not feasible at Visit 3 (Week 2).
Mammography | Week 52 after the surgery
  Mammography will be performed at week 52

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Cardinal Tien Hospital, New Taipei City, Taiwan
  - Taipei Medical University Hospital, Taipei, Taiwan
  - Tri-Service General Hospital, Taipei, Taiwan